CLINICAL TRIAL: NCT06981520
Title: Effect of Caspase-1 Activity, IL-1beta, and IL-18 on Inflammation in the Mucosa of the Small Intestine of Patients With FMF
Brief Title: Caspase-1 Activity, IL-1beta, and IL-18 in Patients With FMF
Acronym: FMF
Status: Not yet recruiting | Type: Observational
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Mustafa Sahin, Principal Investigator, Associate Professor of Medical Biochemistry, Hitit University
Other Study IDs: Hitit University, Çorum; 2025/37 (Other: Hitit University Erol Olçok Training and Research Hospital)
Record Dates: First submitted 2025-04-29; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Familial Mediterranean Fever; Intestinal Disease; Genetic Disease; Fever
MeSH Terms: conditions — Familial Mediterranean Fever; Intestinal Diseases; Genetic Diseases, Inborn; Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples Without DNA — Formalin-fixed paraffin-embedded (FFPE) intestinal mucosal biopsy samples collected during routine endoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup 1: Group Title: FMF Patients Group/Cohort Label: FMF: 1. FMF Patients (Group/Cohort Description) Patients diagnosed with Familial Mediterranean Fever (FMF) according to clinical criteria and/or genetic analysis. Intestinal mucosal biopsy samples were obtained during routine endoscopy, and immunohistochemical staining for IL-1, IL-18, and Caspase-1 was performed.
- Grup 2: Group Title: Healthy Controls Group/Cohort Label: Control: 2. Healthy Controls (Group/Cohort Description) Healthy individuals without any known inflammatory or autoimmune disease, undergoing endoscopy for non-inflammatory indications such as functional gastrointestinal symptoms. Mucosal biopsy samples were collected and analyzed immunohistochemically for IL-1, IL-18, and Caspase-1 expression.

SUMMARY:
This study aims to investigate the intestinal mucosal expression of key inflammatory markers, namely Interleukin-1 (IL-1), Interleukin-18 (IL-18), and Caspase-1, in patients with Familial Mediterranean Fever (FMF). FMF is an autoinflammatory disorder characterized by recurrent episodes of fever and serosal inflammation. Recent studies suggest a possible role of intestinal immune activation in the disease pathogenesis, particularly through inflammasome-related cytokines. To better understand mucosal involvement in FMF, immunohistochemical staining for IL-1, IL-18, and Caspase-1 will be performed on intestinal biopsy samples obtained during routine endoscopic procedures. The staining intensity and distribution patterns will be evaluated and compared with age- and sex-matched healthy controls. The findings may help clarify mucosal inflammatory pathways involved in FMF and provide insight into novel therapeutic targets.

DETAILED DESCRIPTION:
Familial Mediterranean Fever (FMF) is a hereditary autoinflammatory disease characterized by recurrent episodes of fever, serositis, and elevated acute-phase reactants. The underlying pathophysiology involves mutations in the MEFV gene, which encodes pyrin, a protein involved in the regulation of the inflammasome complex. Aberrant inflammasome activation has been associated with increased production of pro-inflammatory cytokines, including interleukin-1 beta (IL-1β) and interleukin-18 (IL-18), mediated through caspase-1 cleavage.

Although FMF primarily affects serosal surfaces, emerging evidence suggests that intestinal mucosal inflammation may also play a role in disease pathogenesis, possibly contributing to atypical symptoms such as abdominal pain, diarrhea, or subclinical intestinal involvement. However, the extent and nature of this mucosal immune activation remain largely unexplored.

This study is designed to evaluate the expression of IL-1, IL-18, and Caspase-1 in intestinal mucosal biopsy specimens obtained from FMF patients during routine endoscopic evaluation. Immunohistochemical staining techniques will be applied to assess the localization and intensity of these markers. The results will be compared to a control group of age- and sex-matched individuals undergoing endoscopy for non-inflammatory indications (e.g., functional gastrointestinal disorders) and without histopathologic mucosal abnormalities.

Staining will be semi-quantitatively scored by two independent pathologists blinded to clinical data. Correlations between cytokine expression levels and clinical characteristics of FMF (e.g., disease duration, mutation status, attack frequency, colchicine response) will also be explored.

This study aims to provide insights into the role of mucosal inflammasome activity in FMF, potentially identifying novel biomarkers or therapeutic targets. By characterizing intestinal expression of key inflammasome-related cytokines, we hope to expand current understanding of FMF pathophysiology beyond classical serosal involvement.

ELIGIBILITY:
Inclusion Criteria:Age 18 years or older

Confirmed diagnosis of Familial Mediterranean Fever (FMF) according to Tel-Hashomer clinical criteria and/or MEFV gene mutation analysis (for FMF group)

Undergoing routine endoscopy with mucosal biopsy sampling

Availability of sufficient formalin-fixed paraffin-embedded (FFPE) tissue for immunohistochemical analysis

For controls: absence of systemic inflammatory or autoimmune disease -

Exclusion Criteria:History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)

Current use of immunosuppressive therapy (excluding colchicine)

Severe infection, active malignancy, or other systemic disease affecting intestinal mucosa

Inadequate biopsy specimen quality for histopathological evaluation

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study includes adult patients diagnosed with Familial Mediterranean Fever (FMF) who underwent routine endoscopic evaluation with intestinal mucosal biopsies. A control group composed of age- and sex-matched individuals without inflammatory or autoimmune diseases was also included for comparative analysis. All participants were retrospectively selected based on availability of adequate tissue samples and relevant clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Level of IL-1 in Mucosal Biopsies (Semi-Quantitative Score) | Single time point, Day 1 (during biopsy analysis)
  Semi-quantitative scoring of immunohistochemical staining in mucosal biopsies; comparison between FMF and control groups
Level of IL-18 in Mucosal Biopsies (Semi-Quantitative Score) | Single time point, Day 1 (during biopsy analysis)
  Semi-quantitative scoring of immunohistochemical staining in mucosal biopsies; comparison between FMF and control groups
Caspase-1 Expression in Mucosal Biopsies (Semi-Quantitative Score) | Single time point, Day 1 (during biopsy analysis)
  Semi-quantitative scoring of immunohistochemical staining in mucosal biopsies; comparison between FMF and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Şahin, Assoc.Prof, Principal Investigator — Hitit University Faculty of Medicine, Turkey
Locations (1):
- Hitit University Erol Olçok Training and Research Hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the retrospective nature and ethical restrictions.